CLINICAL TRIAL: NCT06467396
Title: Blood Biomarkers to Predict the Prognosis of a Stroke Patient Undergoing Mechanical Thrombectomy
Acronym: TROMBOPOCT
Status: Recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Sponsor
Other Study IDs: TROMBOPOCT
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Large Vessel Occlusion Biomarkers Test; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Large Vessel Occlusion Biomarkers Test — Duplex Point of Care test to measure the concentration of blood biomarkers (FABP+NT-proBNP) associated to Large Vessel Occlusion in blood samples used in combination with an APP.

SUMMARY:
The goal of this observational study is to evaluate the accuracy of a panel of blood biomarkers and clinical variables in predicting the prognosis of stroke patients treated by mechanical thrombectomy, specifically to predict futile recanalization and mortality.

DETAILED DESCRIPTION:
Stroke is the leading cause of long-term disability and the second most common cause of death worldwide, accounting for around 6.7 million deaths each year. The burden of stroke due to illness, disability and early death is set to double within the next 15 years due to an ageing population. The socio-economical cost of the stroke is very high, being around 45 million euros per year in Europe. Although mechanical thrombectomy is the most effective treatment for stroke patients with large vessel occlusions still a large percentage of patients, around 50%, do not recover despite a successful recanalization (the so called "futile recanalization"). Therefore, to anticipate the prognosis of patients treated with mechanical thrombectomy would be clinically relevant and very informative.

This observational study evaluates the precision of a rapid test of blood biomarkers in the prognosis of stroke patients treated by mechanical thrombectomy. For that, the investigators will recruit a cohort of 400 consecutive patients treated by thrombectomy. Using a multiplex POC for the biomarker measurement and an APP in combination with clinical data, the potential of biomarkers to predict the prognosis of a patient will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old.
* Patient in whom a mechanical thrombectomy is performed.

Exclusion Criteria:

* Impossibility of getting a blood sample.
* Impossibility of performing the test (Invalid results)
* Refusal to provide the informed consent by the patient/relative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients with large vessel occlusion treated by mechanical thrombectomy
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Specificity and sensibility of blood biomarkers in combination with neurological scales (NIHSS) determined before the thrombectomy intervention to predict the prognosis of the patient (functional dependence and mortality). | through the study completion, an average of one year

SECONDARY OUTCOMES:
Percentage of patients who suffer a futile recanalization after a mechanical thrombectomy. | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen Rocío, Seville